CLINICAL TRIAL: NCT05410483
Title: A Dose-finding Trial of Hyperthermic Intraperitoneal Docetaxel and Cisplatin in Patients Receiving Hyperthermic Intraperitoneal Chemotherapy
Brief Title: A Dose-finding Trial of Hyperthermic Intraperitoneal Docetaxel
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-KY-061
Record Dates: First submitted 2022-05-31; First posted 2022-06-08 (Actual); Last update posted 2022-06-08 (Actual); Status verified 2022-05

CONDITIONS: Hyperthermic Intraperitoneal Chemotherapy
MeSH Terms: interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Docetaxel dose level (Experimental): Initial dose of 60mg/m2 and increase the remaining dose gradient by 5 mg/m2
  Interventions: Drug: Docetaxel

INTERVENTIONS:
Drug: Docetaxel — Hyperthermic Intraperitoneal Docetaxel

SUMMARY:
This is a single-center study design, and 30 patients will be enrolled. Eligible patients will receive docetaxel at different dose levels according to the trial schedule.All the enrolled patients were treated with docetaxel during the first HIPEC treatment and cisplatin during the second HIPEC treatment at 43℃ for 1 hour.The dose of docetaxel for patients in the next group was determined according to the incidence of dose-limiting toxicity (DLT) of the previous docetaxel dose level. Finally, the maximum tolerated dose (MTD) of docetaxel for HIPEC was calculated according to the incidence of dose-limiting toxicity.

DETAILED DESCRIPTION:
This is a single-center study design, and 30 patients will be enrolled. Eligible patients will receive docetaxel at different dose levels according to the trial schedule. All the enrolled patients were treated with docetaxel during the first HIPEC treatment and cisplatin during the second HIPEC treatment at 43℃ for 1 hour. Four dosages of docetaxel were set up in the study. We decided to take the initial dose of 60mg/m2 and increase the remaining dose gradient by 5 mg/m2. The dosage of cisplatin was 75mg/m2. Time-to-event Bayesian Optimal Interval Design(TITE-BOIN) was used, with 3 patients as an observation group (i.e. a cohort), starting from a dose of 60mg/m2. The dose of docetaxel for patients in the next group was determined according to the incidence of dose-limiting toxicity (DLT) of the previous docetaxel dose level. Finally, the maximum tolerated dose (MTD) of docetaxel for HIPEC was calculated according to the incidence of dose-limiting toxicity.

ELIGIBILITY:
Inclusion Criteria:

1. According to the gynecology malignant tumor abdominal hot perfusion chemotherapy clinical expert consensus, with HIPEC treatment indications, including the initial treatment of ovarian cancer, recurrent ovarian cancer, peritoneum pseudo myxoma, accompanied by abdominal cavity effusion or disseminated other gynecological malignant tumors of peritoneal cavity transfer, branch caused by malignant tumors refractory peritoneal effusion, Uterine sarcoma found after the use of tumor (uterine) device, ovarian mucous tumor before or during the rupture, a large amount of mucus overflow contamination of the abdominal cavity.
2. Ages 18 to 70.
3. Serum creatinine was within the normal range (reference range of creatinine: 58-96μmol/L) before receiving HIPEC, and renal function was normal.
4. No bone marrow suppression before HIPEC (considering many factors affecting hemoglobin level, including intraoperative blood loss and postoperative fluid infusion hemodilution, hemoglobin ≥80g/L was set; Leukocyte ≥ 4.0*109/L, granulocyte ≥ 2.0×109/L; Platelet ≥ 100×109/L).
5. No abnormal liver function before receiving HIPEC (total bilirubin 3.4-22.2μmol/L, ALT 7-40 U/L, AST 13-35U/L, AST/ALT≤1.5).
6. Signed informed consent and received docetaxel and cisplatin HIPEC treatment.

Exclusion Criteria:

1. Contraindications to HIPEC: intestinal obstruction; Extensive adhesion in peritoneal cavity; The abdominal cavity has obvious inflammation; There may be high risk factors for poor postoperative anastomotic healing, including anastomotic tissue edema, ischemia, obvious tension, severe hypoproteinemia, etc. Dysfunction of major organs such as heart, kidneys, liver and brain; Severe coagulopathy; Bile obstruction and ureteral obstruction.
2. No history of radiotherapy or chemotherapy in recent 3 weeks.
3. In addition to HIPEC, docetaxel and cisplatin should be used by other means within 3 weeks after HIPEC treatment.
4. Those who have taken drugs that damage liver and kidney function or inhibit bone marrow within 3 months.
5. Allergic to docetaxel and cisplatin.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2023-02-01 (Estimated); Study Completion 2023-02-01 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose of docetaxel | 21 days
  The MTD of docetaxel for abdominal thermal perfusion was calculated by observing the incidence of dose-limiting toxicity 3 weeks after the end of HIPEC.

SECONDARY OUTCOMES:
Incidence of DLT | 9 weeks
  Number of DLT cases at current dose/total cases at current dose
Effect of dose on tumor control rate | 9 weeks
  The decrease of serum CA125 and HE4 concentrations and the results of imaging evaluation at different doses of docetaxel

CONTACTS AND LOCATIONS:
Overall Officials: Zhongqiu Lin, Principal Investigator — Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Locations (1):
- Sun Yat-sen Memorial Hospital, Guangzhou, Other (Non U.s.), China

IPD SHARING:
Plan to Share IPD: No
After data publication

REFERENCES:
- [Derived] You ZY, Wu MF, Li H, Ye YF, Wang LJ, Lin ZQ, Li J. A phase I dose-finding trial of hyperthermic intraperitoneal docetaxel combined with cisplatin in patients with advanced-stage ovarian cancer. J Gynecol Oncol. 2024 Jan;35(1):e1. doi: 10.3802/jgo.2024.35.e1. Epub 2023 Jul 5. PMID 37477105